CLINICAL TRIAL: NCT07167108
Title: "The Effect of the Mulligan Technique on Chronic Neck Pain and Range of Motion in Adults Aged 18 to 65 Years: A Randomized Controlled Trial"
Brief Title: Mulligan Technique for Chronic Neck Pain in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Mosab Saleem Hamed Amoudi (Other)
Responsible Party: Sponsor-Investigator, Prof. Mosab Saleem Hamed Amoudi, Assistant Professor of Physical Therapy, Arab American University (Palestine)
Organization: Arab American University (Palestine) (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAUJ-PT-2025-01
Record Dates: First submitted 2025-08-26; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-03

CONDITIONS: Chronic Neck Pain
Keywords: Neck pain; Mobilization; Mulligan Concept; Mobilization with Movement (MWM); Sustained Natural Apophyseal Glide (SNAG); Range of Motion (ROM)
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group received a conventional physical therapy program (Active Comparator): Control group (A) (n = 32) received a conventional physical therapy program that included exercises, electrical stimulation, and massage.
  Interventions: Other: Conventional Physical Therapy Program
- The experimental group received conventional program, with addition to Mulligan technique (Experimental): The experimental group (B) (n=38) received the same conventional physical therapy program, with the addition of the Mulligan technique.
  Interventions: Other: Conventional program, with addition to Mulligan technique

INTERVENTIONS:
Other: Conventional program, with addition to Mulligan technique — The Mulligan Concept is a manual therapy approach developed by New Zealand physiotherapist Brian Mulligan in the 1980s. It includes techniques such as Mobilization with Movement (MWM) and the Sustained Natural Apophyseal Glide (SNAG), which have attracted significant attention for their effectiveness in treating neck pain. Recent research has supported the benefits of physiotherapy interventions like SNAGs in improving cervical range of motion (ROM) and reducing pain.
  Other Names: Mulligan Concept
  Arms: The experimental group received conventional program, with addition to Mulligan technique
Other: Conventional Physical Therapy Program — Included exercises, electrical stimulation, and massage.
  Arms: Control group received a conventional physical therapy program

SUMMARY:
This study aims to evaluate the effect of the Mulligan Technique, a manual therapy method, on reducing chronic neck pain and improving neck movement in adults aged 18 to 65 years. Participants will receive treatment sessions, and their pain levels and range of motion will be assessed. The goal is to determine if this technique can help improve quality of life for people suffering from chronic neck pain.

DETAILED DESCRIPTION:
Seventy-six participants with chronic neck pain, aged between 18 and 65 years, were selected on the basis of selection criteria. The pain intensity was measured using the Visual Analog Scale (VAS), the cervical range of motion (ROM) was measured using the universal goniometer, and the functional disability was measured using the Neck Disability Index (NDI). Patients were randomly assigned to two Groups A and B. Control group (A) (n = 32) received a conventional physical therapy program that included exercises, electrical stimulation, and massage. The experimental group (B) (n=38) received the same conventional program, with the addition of the Mulligan technique. Six participants were excluded from the study. Both groups underwent treatment 3 times per week for 4 weeks, and measurements were taken before and after the treatment period. For data entry and statistical analysis, (SPSS version 20) was used. The independent samples t-test was capture summarize and interpret data and 95 percent of the confidence interval is covered.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65 years.
* Chronic mechanical neck pain (≥ 3 months).
* Limited cervical range of motion (ROM).
* Medically diagnosed with non-specific neck pain.
* Able to attend treatment sessions.

Exclusion Criteria:

* Radiating pain to the upper limb.
* Signs of nerve root compression or disc herniation.
* History of cervical spine surgery or major trauma.
* Inflammatory joint diseases (e.g., rheumatoid arthritis).
* Osteoporosis or systemic medical conditions affecting bone/joint health.
* Fibromyalgia or central nervous system disorders.
* Contraindications to manual therapy (e.g., pacemaker, vascular disorders).
* Recent physical therapy or steroid injections (within past 3-12 months).
* Long-term use of corticosteroids or pain medications.
* Pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2025-03-02 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pain intensity measured by Visual Analog Scale (VAS) | Before treatment (baseline) and 4 weeks (end of treatment)
  Pain intensity will be measured using a 0-10 Visual Analog Scale at baseline and post-intervention. The change in pain scores will be reported.

SECONDARY OUTCOMES:
Change from baseline in cervical range of motion (ROM) measured by goniometer (degrees) | Before treatment (baseline) and 4 weeks (end of treatment)
  Cervical ROM will be measured in degrees using a goniometer at baseline and post-intervention. The difference between baseline and post-treatment ROM will be reported.
Change from baseline in neck-related disability measured by the Neck Disability Index (NDI) | Before treatment (baseline) and 4 weeks (end of treatment)
  Neck-related disability will be assessed using the Neck Disability Index (NDI), a self-reported questionnaire consisting of 10 items scored on a 0-5 scale. The total score ranges from 0 to 50, with higher scores indicating greater disability. The NDI will be administered at baseline and after the intervention. The change in total NDI score from baseline to post-intervention will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Amoudi, Study Director — Arab American University (Palestine); Mosab S Amoudi, Principal Investigator — Arab American University - Jenin
Locations (1):
- PhysioFlex - Physiotherapy and Rehabilitation Center-Nablus, Nablus, Nablus, Palestinian Territories

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.researchgate.net/profile/Mosab-Amoudi